CLINICAL TRIAL: NCT00340249
Title: Use of a Perinatal Database and Biologic Tissue Bank at the Perinatology Research Branch (PRB)
Brief Title: Use of the Perinatal Database and Biologic Tissue Bank at The Perinatology Research Branch (PRB)
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995040; OH95-CH-N040
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy; Premature Birth; Prenatal Care; Preterm Delivery; Preterm Birth
Keywords: Pregnancy; Preterm Birth; Preterm Birth Prevention; Prematurity; Pregnancy Complications
MeSH Terms: conditions — Premature Birth; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this application is to request permission to use a bank of biological specimens and clinical information collected by the investigators prior to their joining the intramural program. The samples have been gathered under the sponsorship and approval of the Human Investigations Committees at Yale University, Wayne State University and Pennsylvania Hospital in the United States, the Sotero del Rio Hospital, the Hospital of the Universidad de Chile and the Universidad Catolica de Chile , in Chile. The investigators have generated a bank of amniotic fluid, maternal blood and urine, and fetal blood obtained at the time of delivery (from the umbilical cord and by cordocentesis), neonate s urine and sonographic examinations of the fetus, including echocardiography, stored on videotapes. Clinical information with patient identifiers is available for these samples and sonographic examinations.

DETAILED DESCRIPTION:
The purpose of this application is to request permission to use a bank of biological specimens and clinical information collected by the investigators prior to their joining the intramural program. The samples have been gathered under the sponsorship and approval of the Human Investigations Committees at Yale University, Wayne State University and Pennsylvania Hospital in the United States, the Sotero del Rio Hospital, the Hospital of the Universidad de Chile and the Universidad Catolica de Chile , in Chile. The investigators have generated a bank of amniotic fluid, maternal blood and urine, and fetal blood obtained at the time of delivery (from the umbilical cord and by cordocentesis), neonate s urine and sonographic examinations of the fetus, including echocardiography, stored on videotapes. Clinical information with patient identifiers is available for these samples and sonographic examinations.

ELIGIBILITY:
* Not listed in protocol - samples only.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20964 (Actual)
Dates: Start 1995-08-22 (Actual); Primary Completion 2007-09-18 (Actual); Study Completion 2007-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Krebs C, Macara LM, Leiser R, Bowman AW, Greer IA, Kingdom JC. Intrauterine growth restriction with absent end-diastolic flow velocity in the umbilical artery is associated with maldevelopment of the placental terminal villous tree. Am J Obstet Gynecol. 1996 Dec;175(6):1534-42. doi: 10.1016/s0002-9378(96)70103-5. PMID 8987938
- [Background] Baker PN, Krasnow J, Roberts JM, Yeo KT. Elevated serum levels of vascular endothelial growth factor in patients with preeclampsia. Obstet Gynecol. 1995 Nov;86(5):815-21. doi: 10.1016/0029-7844(95)00259-T. PMID 7566855
- [Background] Torry DS, Wang HS, Wang TH, Caudle MR, Torry RJ. Preeclampsia is associated with reduced serum levels of placenta growth factor. Am J Obstet Gynecol. 1998 Dec;179(6 Pt 1):1539-44. doi: 10.1016/s0002-9378(98)70021-3. PMID 9855593